CLINICAL TRIAL: NCT03320525
Title: A Single Center, Open-Label, Phase 1 Study to Evaluate the Pharmacokinetic Profile of T-ChOS™ in Subjects With Advanced Solid Tumors (CHITIN)
Brief Title: Pharmacokinetic Profile of T-ChOS™ in Subjects With Advanced Solid Tumors (CHITIN)
Acronym: CHITIN
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues with PK detection limits and compliance to protocol at the analytical site.
Sponsor: Herlev Hospital (Other)
Collaborators: GENIS (Unknown)
Responsible Party: Principal Investigator, Inna Chen, MD, Principal Investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA1602
Record Dates: First submitted 2017-10-14; First posted 2017-10-25 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Advanced Solid Tumors
Keywords: YKL-40; Pharmacokinetic; Solid tumors; T-ChOS; Benecta; chitinase 3 like-1 protein (CHI3L1)

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The active substance used in the T-ChOS capsule formulation is a chitooligosaccharide blend.
  Interventions: Dietary Supplement: T-ChOS

INTERVENTIONS:
Dietary Supplement: T-ChOS — T-ChOS 600 mg (two capsules, each 300 mg) daily in the morning 30 minutes before food.

SUMMARY:
This is a single center phase 1 trial, which evaluates the pharmacokinetic profile of T-ChOS™ (food supplement Benecta™) in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
YKL-40 (also named chitinase 3 like-1 protein, CHI3L1), is a member of the mammalian chitinase like proteins and is a highly conserved glycoprotein. YKL-40 is produced by cancer cells and macrophages and promotes cancer progression by activating inflammation and inhibiting tumor angiogenesis. Thus, YKL-40 could be a new therapeutic target for patients with cancer.

T-ChOS™ is a technical name for a food supplement product that is marketed in Iceland under the name Benecta™. T-ChOS is manufactured using shellfish derived chitin as a raw material and is produced by Genis in Iceland. It is a blend of chitooligosaccharides that are hetero-complexes of N-acetyl-glucosamine and D-glucosamine. T-ChOS chitooligosaccharides have been specially selected to have high bioactivity in inflammatory models and strong binding affinity to YKL-40. Chitooligosaccharide induced blockade of YKL-40 signalling pathways may represents a promising approach. Pharmacokinetic profile of the T-ChOS in patients with advanced solid malignancies is not available.

Safety and tolerability data will be collected to expand the safety/tolerability database for patients with advanced solid malignancies treated with oral T-ChOS. Patients will be allowed to receive T-ChOS on a continuous basis and therefore have the possibility to gain clinical benefit, if any. Safety and tolerability data collected after pharmacokinetic part of the study will be also added to the safety database for patients with advanced solid malignancies treated with oral T-ChOS.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed written Informed Consent
* Male or females aged 18 to 75 years at the time of signing the informed consent form (ICF)
* Patients must have histological confirmed malignancy (solid tumor) that is metastatic or unresectable and for which standard curative or palliative therapies do not exist or are no longer effective
* Understand and voluntarily sign an ICF prior to any study related assessments or procedures being conducted
* Performance status 0-1 (ECOG)
* Life expectancy ≥ 3 months
* Elevated blood YKL-40 > 40 μg/L, assessed within 28 days prior to the start of the study
* Hematopoietic

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Platelet count ≥ 100 x 10⁹/L
  * Haemoglobin ≥ 5.6 mmol/L
* Hepatic

  * Serum bilirubin < 1.5 x upper limit of normal (ULN)
  * AST/ALT < 2.5 x ULN (< 5 x ULN with known liver metastasis)
* Renal

  * Acceptable renal function with a creatinine clearance ≥ 50 mL/min/ (e.g., using the Cockroft-Gault formula)
* Cardiovascular

  * No severe or uncontrolled cardiac condition
* Pulmonary

  * No severe or uncontrolled pulmonary condition
* Immunologic

  * No known or suspected allergy to the investigational product
* Gastrointestinal

  * No chronic enteropathy (e.g. active inflammatory bowel disease, extensive intestinal resection or chronic diarrhea)
  * No bowel obstruction or sub-obstruction
  * No prior history of intestinal malabsorption
  * Patients have to be able to swallow normally and have to be willing to comply with the intake of capsules
* Others

  * No psychiatric condition that would preclude study participation
  * No co-existing active infection requiring antibiotics or any co-existing medical conditions likely to interfere with study procedures
  * No other condition that will preclude study participation
  * A negative pregnancy test for women of childbearing potential. For men and women of child-producing potential, the use of effective contraceptives methods during the study and at least 3 months after discontinuations of the investigational product is required. The following contraceptive methods are regarded as effective: intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release). Sterilised or infertile patients are exempt from the requirement to use contraception. In order to be considered sterilised or infertile, patients must generally have undergone surgical sterilisation (vasectomy/bilateral tubectomy, hysterectomy or bilateral ovariectomy) or be postmenopausal defined as 12 months or more with no menses prior to enrolment
  * Not pregnant or nursing
* Be able to adhere to the study visit schedule and other protocol requirements

EXCLUSION CRITERIA:

* Simultaneous participation in any other study involving investigational drugs or having participated in a study within 2 weeks prior to start of study treatment
* Current use of anticoagulation therapy such as heparins both unfractionated and low molecular weighted
* Symptomatic brain metastases
* Intake of any prohibited concomitant medication
* Prior and Concurrent Therapy at least 2 weeks prior to 1st dosing:

  * Biologic/immunotherapy
  * Chemotherapy
  * Radiotherapy
  * Major or laparoscopic surgery
  * Other concurrent anticancer therapy
  * Corticosteroids or other immunosuppressive medications. Inhaled or topical steroids are permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters will be assessed for T-ChOS | Approximately up to 12 months
  • time to reach maximum plasma concentration (tmax)
Pharmacokinetic parameters will be assessed for T-ChOS | Approximately up to 12 months
  • area under the plasma concentration-time curve from zero to the last measurable time point (AUC0-t)
Pharmacokinetic parameters will be assessed for T-ChOS | Approximately up to 12 months
  • area under the plasma concentration-time curve from zero to infinity (AUC)
Pharmacokinetic parameters will be assessed for T-ChOS | Approximately up to 12 months
  • apparent plasma clearance following oral administration (CL/F)
Pharmacokinetic parameters will be assessed for T-ChOS | Approximately up to 12 months
  • terminal half-life (t½)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Approximately up to 18 months.
  Safety and tolerability of the treatment regimens assessed by a summary of adverse events and clinical laboratory assessments.
Overall response rate (ORR) | Approximately up to 18 months.
  ORR = complete response + partial response, according to RECIST 1.1
Disease control rate (DCR) | Approximately up to 18 months.
  DCR = complete response + partial response + stable disease, according to RECIST 1.1

OTHER OUTCOMES:
Serum YKL-40 | Approximately up to 18 months.
  Serum YKL-40 during and following 4 weeks of treatment with T-ChOS
Serum CRP | Approximately up to 18 months.
  Serum CRP during and following 4 weeks of treatment with T-ChOS

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark